CLINICAL TRIAL: NCT06066060
Title: Phase I Study to Evaluate the Drug-Drug Interaction (DDI) Between JMKX000623 Tablets and Metformin Hydrochloride Tablets in Healthy Chinese Subjects
Brief Title: A DDI Study of JMKX000623 and Metformin Hydrochloride
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jemincare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: JY-JM025-102
Record Dates: First submitted 2023-09-13; First posted 2023-10-04 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Healthy; Drug-Drug Interaction
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JMKX000623/Metformin/ JMKX000623+Metformin (Experimental): D1-D8, JMKX000623; D14-D19, Metformin; D20-D27, JMKX000623+Metformin
  Interventions: Drug: JMKX000623; Drug: Metformin

INTERVENTIONS:
Drug: JMKX000623 — JMKX000623, administered orally ;
Drug: Metformin — Metformin,administered orally

SUMMARY:
A phase 1, single center, 1 sequence, 3 period, open label, multiple doses study to evaluate the drug-drug interaction of JMKX000623 tablet and metformin.

DETAILED DESCRIPTION:
The drug-drug interaction study is meant to evaluate the pharmacokinetics and safety of JMKX000623 tablet combined metformin in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Chinese subjects aged 18-45 years, male or female;
2. Weight: male≥50.0kg, female≥45.0kg, 19.0 kg/m2≤BMI<27.0 kg/m2;
3. Normal or abnormal but without clinical significance reports of physical examinations, vital signs, clinical laboratory tests and others;
4. Able to provide written informed consent voluntarily.

Exclusion Criteria:

1. Suspected hypersensitivity to the main ingredients and excipients of JMKX000623 tablets, metformin hydrochloride tablets, or a history of allergy to drugs, food or other substances;
2. History of clinically significant chronic gastrointestinal disease or history of gastrointestinal surgery (excluding appendectomy) that the investigator believes may affect drug absorption;
3. Surgery within 3 months prior to screening that, in the judgment of the investigator, would interfere with the absorption, distribution, metabolism, or excretion of the drug, or surgery within 4 weeks prior to the use of the investigational drug, or planned surgery during the research;
4. Took any prescription, over-the-counter, and herbal medications within 2 weeks prior to screening, or were within 5 half-lives of the medication at the time of screening, and plan to take other experimental medications other than those in this study for the duration of the research;
5. Other conditions unsuitable for the study confirmed by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-09-17 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-11-06 (Actual)

PRIMARY OUTCOMES:
Area Under the Dosing Time Curve During the Dosing Interval After Reaching Steady State（AUC0-tau） | baseline through 4 days post-dose
Maximum observed After Reaching steady state concentration (Css,max) | baseline through 4 days post-dose

SECONDARY OUTCOMES:
Adverse events (AEs) | baseline through 4 days post-dose
  Incidence and features of AEs assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojie Wu, MD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No